CLINICAL TRIAL: NCT06465680
Title: Intern Health Study: 2024 Cohort Micro-Randomized Trial
Brief Title: Intern Health Study 2024
Acronym: IHS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Srijan Sen, Research Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH-101459-2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Depression; Mood; Sleep; Physical Activity
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-participant micro-randomization (Experimental): Each day in the study, with probability .5 for each, a participant is randomized to receive a notification that day or no notification that day.
  If a participant is assigned to receive a notification that day, 1 message set will be randomly selected from a pool of 358 core message sets. Each core message set will be comprised of 4 messages containing comparable content, however they will be tailored based on the participant's wearable (steps, sleep) or mood data for the specified time interval (7 days, 30 days, since the start of internship) as follows: 1) no data, 2) low, 3) moderate, or 4) high.
  Interventions: Behavioral: Intern Health Study behavioral change mobile notification

INTERVENTIONS:
Behavioral: Intern Health Study behavioral change mobile notification — The study's mobile app will be used to deliver push notifications. The notifications appear on the participant's phone lock screen. The notifications include 3 categories: mood notifications, activity notifications, sleep notifications. Mood notifications aim to increase the participant's mood. Activity notifications aim to increase the participant's physical activity. Sleep notifications aim to increase the participant's sleep duration. All notifications are categorized as one of five therapeutic approaches: 1) CBT-Behavioral, 2) CBT-Cognitive, 3) Distanced Self-Talk, 4) Mindfulness, 5) Motivational Interviewing.

SUMMARY:
The aim of this trial is to evaluate the efficacy of an intervention (delivered through a smartphone) for improving the mood, physical activity, and sleep of medical interns.

DETAILED DESCRIPTION:
Due to their high stress workloads, medical interns suffer from depression at higher rates than the general population. Interns also tend to have lower sleep and decreased physical activity. The goal of this trial is to evaluate the efficacy of a mobile health intervention intending to help improve the mental health of medical interns. The intervention sends mobile phone notifications which aim to help interns improve their mood, maintain physical activity, and obtain adequate sleep during their internship year.

The primary aim of the study is to evaluate how notifications affect participants' weekly mood, as measured through a daily one question mood survey. The second primary aim of the study is to evaluate how notifications affect participants' long-term mental health, as measured by the Patient Health Questionnaire. The first secondary aim is to evaluate how mood notifications affect participants' weekly mood. The second secondary aim is to evaluate how activity notifications affect participants' weekly step count. The third secondary aim is to evaluate how sleep notifications affect participants' weekly sleep duration. In order to better optimize notification delivery, the final aim (exploratory) is to understand moderators of these effects. Moderators of interest are previous week's mood, previous week's step count, previous week's sleep duration, study week, sex, previous history of depression, and baseline neuroticism.

ELIGIBILITY:
Inclusion Criteria:

* Medical intern during the 2024-2025 internship year
* iPhone or Android phone user
* Logged into the Intern Health Study mobile app, completed consent, and filled out baseline survey by June 30 prior to the start of intern year

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Average daily mood | Daily, through study completion at the end of intern year (1 year)
  Through the mobile app, participants enter a mood score (scale 1 - 10) every day of the study. 1 corresponds to lowest mood and 10 corresponds to highest mood.
Average daily step count | Daily, through study completion at the end of intern year (1 year)
  Participant's daily step counts are recorded through a fitness tracker. High step counts are considered a positive outcome as it indicates more physical activity.
Average nightly sleep duration | Daily, through study completion at the end of intern year (1 year)
  Participant's nightly sleep duration (in minutes) is recorded through a fitness tracker. High sleep duration is considered a positive outcome.
Patient Health Questionnaire-9 (PHQ-9) | Quarterly (every 3 months for 1 year)
  Prior to the start of the intervention and at quarterly intervals throughout internship year, all participants complete the Patient Health Questionnaire 9. High scores on the PHQ-9 correspond to a larger number of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified genomic and survey information (baseline survey, plus quarterly survey which contains the PHQ-9) will be shared with the National Institute for Mental Health (NIMH).
Supporting Information: ICF
Time Frame: Data will be made available 12 months after the end of the trial. It will be made available indefinitely after that date.
Access Criteria: The data will be shared directly with the NIMH. NIMH will apply their criteria for qualified researchers and analyses.
URL: https://www.openicpsr.org/openicpsr/project/129225/version/V1/view

REFERENCES:
- See also: Sen Lab Website — https://www.srijan-sen-lab.com/intern-health-study
- See also: Study Participant Website — https://www.internhealthstudy.org/